CLINICAL TRIAL: NCT01029548
Title: Observational Study With Additional Diagnostic Procedures on Anti-Tat Immune Response in HIV-1-infected Asymptomatic Adult Subjects
Brief Title: Observational Study on Anti-Tat Immune Response in HIV-1-infected Asymptomatic Adult Subjects
Acronym: ISS OBS T-003
Status: Completed | Type: Observational
Sponsor: Barbara Ensoli, MD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS OBS T-003
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: HIV; Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, serum, PBMCs
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed as a prospective observational study directed at evaluating the frequency, magnitude, quality and persistence (primary endpoint) of the anti-Tat immune response in HIV-1 infected asymptomatic individuals, and to prospectively evaluate the immunological, virological and clinical outcome of anti-Tat positive versus anti-Tat negative drug naїve subjects (secondary endpoint) in order to determine the impact of anti-Tat immunity on HIV disease progression as well as the potential use of anti-Tat immune response assessment for the clinical and therapeutic management of infected patients. This survey provided important information for the design, planning and conduction of future therapeutic vaccine trials based on the HIV-1 Tat protein in asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

* To be clinically asymptomatic HIV-1 infected individuals with CD4+ T cell counts ≥400/μL
* To be naïve for antiretroviral therapy
* Levels of plasma viremia ≤100,000 copies/ml at baseline
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Current therapy with immunomodulators or immunosuppressive drugs or chemotherapy for neoplastic disorders
* Concomitant treatment for HBV or HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic HIV infected individuals
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2008-04; Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Specific humoral and cellular immune responses to Tat will be monitored by assessing anti-Tat specific antibodies in sera, proliferative response (CFSE) and production of γIFN, IL-4 and IL-2 (Elispot) by peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
The decline of CD4+ T cells count, the increase of the HIV plasma viral load or the occurrence of AIDS-defining events will be assessed to determine the progression to disease

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mazzotta, MD, Principal Investigator — A.M. Annunziata Hospital Florence, Italy; Giuseppe Pastore, MD, Principal Investigator — General Hospital of Bari; Florio Ghinelli, MD, Principal Investigator — General Hospital-University of Ferrara; Roberto Esposito, MD, Principal Investigator — General Hospital-University of Modena; Massimo Galli, MD, Principal Investigator — L.Sacco Hospital - MI; Fabrizio Soscia, MD, Principal Investigator — S.M. Goretti Hospital Latina; Guido Palamara, MD, Principal Investigator — San Gallicano Hospital - Rome; Adriano Lazzarin, MD, Principal Investigator — San Raffaele Hospital - Milan; Giampiero Carosi, MD, Principal Investigator — Spedali Civili - Brescia; Giovanni Di Perri, MD, Principal Investigator — Amedeo di Savoia Hospital - Turin
Locations (10):
- Italy (10):
  - Giovanni Di Perri, Turin, Italy
  - S.M. Goretti Hospital, Latina, Rome
  - General Hospital of Bari, Bari
  - Spedali Civili di Brescia, Brescia
  - General Hospital-University of Ferrara, Ferrara
  - A.M. Annunziata Hospital, Florence
  - L. Sacco Hospital, Milan
  - San Raffaele Hospital, Milan
  - General Hospital-University of Modena, Modena
  - San Gallicano Hospital, Rome

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Rodman TC, To SE, Hashish H, Manchester K. Epitopes for natural antibodies of human immunodeficiency virus (HIV)-negative (normal) and HIV-positive sera are coincident with two key functional sequences of HIV Tat protein. Proc Natl Acad Sci U S A. 1993 Aug 15;90(16):7719-23. doi: 10.1073/pnas.90.16.7719. PMID 7689227
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Result] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- See also: Related Info — http://www.hiv1tat-vaccines.info